CLINICAL TRIAL: NCT01850420
Title: A Double-Blinded, Randomized, Placebo-Controlled, Proof of Concept Phase 2a Study Exploring the Safety and Efficacy of IMC-1 for the Treatment of Patients With Fibromyalgia
Brief Title: A Study of IMC-1 In Patients With Fibromyalgia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Innovative Med Concepts, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PRID-201
Record Dates: First submitted 2013-05-07; First posted 2013-05-09 (Estimated); Last update posted 2015-03-27 (Estimated); Status verified 2015-03

CONDITIONS: Fibromyalgia; Chronic Pain; Myofascial Pain
Keywords: fibromyalgia; Myofascial
MeSH Terms: conditions — Fibromyalgia; Chronic Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- IMC-1 (Experimental): Experimental intervention
  Interventions: Drug: IMC-1
- Matching placebo (Placebo Comparator)

INTERVENTIONS:
Drug: IMC-1
  Arms: IMC-1

SUMMARY:
This is a randomized, double-blind, placebo-controlled, 16-week study designed to evaluate the hypothesis that tissue-resident herpes virus may be causally related to fibromyalgia symptoms or recurrence. IMC-1 is a combination treatment that is designed to suppress this suspected virus and thus alleviate fibromyalgia symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of fibromyalgia
* English speaker

Exclusion Criteria:

* Rheumatologic diseases
* Bipolar disease, OCD, severe anxiety, schizophrenia
* Systemic infection, severe cardiac disease, chronic steroid usage
* chronic opioid usage

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2013-05; Primary Completion 2014-01 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Change in pain from baseline | 16 weeks
  Comparison of the change from baseline in patient self reported pain scores between IMC-1 and placebo treatment, over 16 weeks of treatment

SECONDARY OUTCOMES:
Patient Global Impression of Change | 16 weeks
  Patients will rate their global improvement over the duration of the trial
Fibromyalgia Impact Questionnaire | 16 weeks

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - IMC Study Site, Birmingham, Alabama
  - IMC Study Site, Sacramento, California
  - IMC Study Site, San Diego, California
  - IMC Study Site, Vista, California
  - IMC Study Site, Jacksonville, Florida
  - IMC Study Site, Tampa, Florida
  - IMC Study Site, Evansville, Indiana
  - IMC Study Site, Lafayette, Indiana
  - IMC Study Site, Ann Arbor, Michigan
  - IMC Study Site, Raleigh, North Carolina
  - IMC Study Site, Medford, Oregon
  - IMC Study Site, Salt Lake City, Utah